CLINICAL TRIAL: NCT01616745
Title: Characteristics of Patients With Nontuberculosis Mycobacteria in Korean Population
Brief Title: Phenotypic Clinical, and Genetic Characteristics of Patients With Nontuberculosis Mycobacteria
Acronym: Korean NTM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Joon Yim, Professor, Seoul National University Hospital
Other Study IDs: H-1103-057-355
Record Dates: First submitted 2012-03-25; First posted 2012-06-12 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Nontuberculosis Mycobacterial Lung Disease
Keywords: NTM Lung disease; NTM Lung disease patients enrolled in SNUH

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to elucidate phenotypic, clinical, and genetic characteristics of Korean Nontuberculosis Mycobacteria (NTM) patients.

DETAILED DESCRIPTION:
To elucidate phenotypic, clinical, and genetic characteristics of Korean NTM patients.

Especially, to compare body mass index, positive rate of IGRA, and CFTR mutation with general Korean population.

ELIGIBILITY:
Inclusion Criteria:

* Persons met diagnostic criteria of NTM lung disease by ATS/IDSA on 2007

Exclusion Criteria:

* Already on treatment for NTM lung disease
* Appropriate exclusion of other lung diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: persons met diagnostic criteria of NTM lung disease by ATS/IDSA on 2007
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-07; Study Completion 2021-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Joon Yim, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Hyung K, Kim SA, Kwak N, Yim JJ, Kim JY. Clinically significant hemoptysis and all-cause mortality in patients with nontuberculous mycobacterial pulmonary disease. Respir Med. 2025 Feb;237:107946. doi: 10.1016/j.rmed.2025.107946. Epub 2025 Jan 8. PMID 39793860
- [Derived] Hyung K, Kim SA, Kim JY, Kwak N, Yim JJ. Rates and Risk Factors of Progression in Patients With Nontuberculous Mycobacterial Pulmonary Disease: Secondary Analysis of a Prospective Cohort Study. Chest. 2024 Sep;166(3):452-460. doi: 10.1016/j.chest.2024.03.024. Epub 2024 Mar 16. PMID 38499238
- [Derived] Kwak N, Park J, Kim SJ, Kim JY, Kim TS, Yoon JK, Whang J, Lee W, Shin SJ, Yim JJ. Genetic stability of Mycobacterium abscessus during antibiotic treatment. J Glob Antimicrob Resist. 2024 Mar;36:45-49. doi: 10.1016/j.jgar.2023.12.004. Epub 2023 Dec 19. PMID 38128724
- [Derived] Jung HI, Kim SA, Kim HJ, Yim JJ, Kwak N. Anxiety and Depression in Patients With Nontuberculous Mycobacterial Pulmonary Disease: A Prospective Cohort Study in South Korea. Chest. 2022 Apr;161(4):918-926. doi: 10.1016/j.chest.2021.10.024. Epub 2021 Oct 28. PMID 34756943
- [Derived] Kwak N, Lee JH, Kim HJ, Kim SA, Yim JJ. New-onset nontuberculous mycobacterial pulmonary disease in bronchiectasis: tracking the clinical and radiographic changes. BMC Pulm Med. 2020 Nov 10;20(1):293. doi: 10.1186/s12890-020-01331-3. PMID 33172424
- [Derived] Kwak N, Whang J, Yang JS, Kim TS, Kim SA, Yim JJ. Minimal Inhibitory Concentration of Clofazimine Among Clinical Isolates of Nontuberculous Mycobacteria and Its Impact on Treatment Outcome. Chest. 2021 Feb;159(2):517-523. doi: 10.1016/j.chest.2020.07.040. Epub 2020 Jul 24. PMID 32712225
- [Derived] Kwak N, Kim SA, Choi SM, Lee J, Lee CH, Yim JJ. Longitudinal changes in health-related quality of life according to clinical course among patients with non-tuberculous mycobacterial pulmonary disease: a prospective cohort study. BMC Pulm Med. 2020 May 7;20(1):126. doi: 10.1186/s12890-020-1165-3. PMID 32381080
- [Derived] Kim HJ, Lee JH, Yoon SH, Kim SA, Kim MS, Choi SM, Lee J, Lee CH, Han SK, Yim JJ. Nontuberculous mycobacterial pulmonary disease diagnosed by two methods: a prospective cohort study. BMC Infect Dis. 2019 May 24;19(1):468. doi: 10.1186/s12879-019-4078-0. PMID 31126235
- [Derived] Kim SJ, Yoon SH, Choi SM, Lee J, Lee CH, Han SK, Yim JJ. Characteristics associated with progression in patients with of nontuberculous mycobacterial lung disease : a prospective cohort study. BMC Pulm Med. 2017 Jan 5;17(1):5. doi: 10.1186/s12890-016-0349-3. PMID 28056937
- [Derived] Lee AR, Lee J, Choi SM, Seong MW, Kim SA, Kim M, Chae KO, Lee JS, Yim JJ. Phenotypic, immunologic, and clinical characteristics of patients with nontuberculous mycobacterial lung disease in Korea. BMC Infect Dis. 2013 Nov 25;13:558. doi: 10.1186/1471-2334-13-558. PMID 24274658